CLINICAL TRIAL: NCT00890617
Title: A Pilot Study of Percutaneous Cryotherapy as Treatment for Stage I Lung Cancer or Solitary Metastatic Lung Cancer
Brief Title: Cryotherapy in Treating Patients With Primary Stage I Non-Small Cell Lung Cancer or Lung Metastasis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frank Baciewicz Jr., Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-048; P30CA022453 (NIH); WSU-2008-048
Record Dates: First submitted 2009-04-29; First posted 2009-04-30 (Estimated); Results first posted 2020-07-29 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Lung Cancer; Metastatic Cancer
Keywords: lung metastases; stage I non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplasm Metastasis; Carcinoma, Non-Small-Cell Lung | interventions — Cryotherapy; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Prednisone & Cryotherapy (Experimental): Prednisone taken:
  20mg BID on the day of the cryotherapy procedure 20mg BID on the day after the procedure 20mg BID two days after the procedure 20mg AM and 10mg PM three days after the procedure 10mg AM and 10mg PM four days after the procedure 10mg five days after the procedure 5mg six days after the procedure
  Interventions: Procedure: Cryotherapy (PTC); Drug: Prednisone

INTERVENTIONS:
Procedure: Cryotherapy (PTC) — CT-guided PTC with the intent to eradicate the entire tumor(s).
Drug: Prednisone — Prednisone taken:
  20mg BID on the day of the cryotherapy procedure 20mg BID on the day after the procedure 20mg BID two days after the procedure 20mg AM and 10mg PM three days after the procedure 10mg AM and 10mg PM four days after the procedure 10mg five days after the procedure 5mg six days after the procedure
  Other Names: Rayos; Sterapred

SUMMARY:
RATIONALE: Cryotherapy kills tumor cells by freezing them. Giving cryotherapy before surgery may kill more tumor cells.

PURPOSE: This phase I trial is studying how well cryotherapy works in treating patients with primary stage I non-small cell lung cancer or lung metastasis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Evaluate the histologic result of treating patients with primary stage I non-small cell lung cancer or lung metastasis after neoadjuvant percutaneous cryotherapy (PTC).

Secondary

* Provide a qualitative assessment of the histology from the ablation and tumor margins, comparing histologic observations with imaging-enhancement patterns by CT or PET scan before and after PTC.

OUTLINE: Patients undergo CT-guided percutaneous cryotherapy (PTC) over 2 hours. Approximately 3 weeks after completion of PTC, patients undergo thoracotomy consisting of lobectomy of the primary lung cancer or wedge resection with adequate margin for the metastatic lesion, and mediastinal lymph node dissection.

Tissue samples from ablation and tumor margins are collected during thoracotomy and compared with imaging-enhanced patterns of CT or PET scans taken at baseline and after PTC.

After completion of study therapy, patients are followed periodically for 6 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed (by percutaneous transthoracic needle biopsy or transbronchial biopsy) diagnosis of 1 the following:

  * Non-small cell lung carcinoma

    * Stage I disease
    * Primary disease
    * No primary lung metastatic disease, satellite lesions of the chest, mediastinal lymph nodes > 1.5 cm, hepatic or adrenal masses by the PET scan or the CT scan
  * Metastatic cancer to the lung

    * Must have a definitive cancer diagnosis with the primary tumor under local control and no metastatic disease other than to the lung
    * Solitary or multiple (≤ 3) peripheral lung lesions
    * No chemotherapy since the new metastatic lesion appeared
* Measurable disease, defined as 1 lesion unidimensionally measured ≤ 3.0 cm by conventional CT scan techniques
* Must be registered with the Clinical Trials office at the Karmanos Cancer Center/Wayne State University
* Must be a candidate for a thoracotomy
* No evidence of cerebral disease or metastatic disease of the brain

PATIENT CHARACTERISTICS:

* Neutrophil count > 1,500/mm^3
* Platelet count > 75,000/mm^3
* PT and PTT normal
* FEV_1 > 1.0 L/sec
* Diffusing capacity ≥ 30%
* Not pregnant or nursing
* No other uncontrolled or concurrent illnesses including, but not limited to, any of the following conditions:

  * Active infection
  * Heart failure
  * Unstable angina
  * Cardiac dysrhythmia
  * Psychiatric illness or a social situation that would limit compliance with the study requirements

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior radiation therapy or chemotherapy for these particular tumors
* No concurrent aspirin or other platelet-inhibiting drugs (e.g., coumadin or heparin)
* No other concurrent experimental studies

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2009-03; Primary Completion 2019-07-27 (Actual); Study Completion 2021-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank A. Baciewicz, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

REFERENCES:
- See also: Clinical trial summary from the National Cancer Institute's PDQ® database — http://cancer.gov/clinicaltrials

RESULTS

PARTICIPANT FLOW:
Groups:
- Prednisone & Cryotherapy: Prednisone taken:
  20mg BID on the day of the cryotherapy procedure 20mg BID on the day after the procedure 20mg BID two days after the procedure 20mg AM and 10mg PM three days after the procedure 10mg AM and 10mg PM four days after the procedure 10mg five days after the procedure 5mg six days after the procedure
  Cryotherapy (PTC): CT-guided PTC with the intent to eradicate the entire tumor(s).
  Prednisone: Prednisone taken:
  20mg BID on the day of the cryotherapy procedure 20mg BID on the day after the procedure 20mg BID two days after the procedure 20mg AM and 10mg PM three days after the procedure 10mg AM and 10mg PM four days after the procedure 10mg five days after the procedure 5mg six days after the procedure
Period: Overall Study
Arm/Group | Prednisone & Cryotherapy
Started | 9
Completed | 9
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prednisone & Cryotherapy
Number analyzed (Participants) | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 5
Age, Continuous [Mean (Full Range); unit: years] | 65.78 [52 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 9

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With a Response (Complete Response and Partial Response)
Description: Treatment success was defined as > 75% of the resected ablated tissue showing no cancer on detailed histologic analysis. The primary statistical objective was to estimate the PCA success rate (p).
Time Frame: 3 weeks post-Percutaneous Cryotherapy (PTC)
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone & Cryotherapy
Number analyzed (Participants) | 9
Participants | 8

2. Secondary Outcome: The Number of Patients With a Pathologic Response
Description: Histology samples from anterior, posterior, superior, inferior, medial and lateral areas of the resected tumor will be compared to enhancement zones of the ablation margin for any residual cancer.
Time Frame: 6 months post-Percutaneous Cryotherapy (PTC)
Measure: Count of Participants; unit: Participants
Arm/Group | Prednisone & Cryotherapy
Number analyzed (Participants) | 9
Participants
  macroscopic residual viable tumor | 1
  microscopic foci of viable tumor | 2
  no microscopic viable tumor | 6

ADVERSE EVENTS:
Time Frame: over the first 6 months of study
Description: CTCAE criteria
Arm/Group | Prednisone & Cryotherapy
All-Cause Mortality (participants affected / at risk) | 2/9
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone & Cryotherapy (N=9)
aspergillosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
atrial fibrillation (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prednisone & Cryotherapy (N=9)
atrial fibrillation (Cardiac disorders) | 2 (2)
pneumonia (Infections and infestations) | 2 (2)
atelectasis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
vocal cord dysfunction (Injury, poisoning and procedural complications) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2012-05-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT00890617/Prot_SAP_000.pdf